CLINICAL TRIAL: NCT06203613
Title: Clinical Study of CLDN18.2 PET/CT for Noninvasive Diagnosis of Gastric and Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: YiHui Guan (Other)
Responsible Party: Sponsor-Investigator, YiHui Guan, Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-1015
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Positron Emission Tomography; Pancreatic Neoplasms; Igestive System Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with gastric cancer (Experimental): Subjects were recruited from the Department of General Surgery, Huashan Hospital, Fudan University, Shanghai, China.
  Interventions: Radiation: [18F]F-H3RESCA-3A12及[68Ga]Ga-NOTA-3A12
- patients with pancreatic cancer (Experimental): Subjects were recruited from the Department of General Surgery, Huashan Hospital, Fudan University, Shanghai, China.
  Interventions: Radiation: [18F]F-H3RESCA-3A12及[68Ga]Ga-NOTA-3A12

INTERVENTIONS:
Radiation: [18F]F-H3RESCA-3A12及[68Ga]Ga-NOTA-3A12 — The dose of [18F]RCCB6 was calculated based on the patient's body weight to be 3.7 MBq [0.1 MCi]/kg, and the method of administration was intravenous push, with a single visualization administered once.

SUMMARY:
In this study, we will investigate the diagnostic efficacy and safety of [18F]F-H3RESCA-3A12 and [68Ga]Ga-NOTA-3A12 in metastatic gastric and pancreatic cancers, and evaluate the sensitivity and specificity of the use of [18F]F-H3RESCA-3A12 and [68Ga]Ga-NOTA-3A12 for diagnosing metastatic gastric and pancreatic cancers . This study will provide a new method for the noninvasive target-specific diagnosis of gastric and pancreatic cancer, and provide intuitive and clear imaging basis for clinical diagnosis, differential diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age between 18 and 65 years old, gender is not limited. (2) Patients with gastric or pancreatic cancer confirmed by puncture or surgical pathology.

  (3) Written informed consent signed by the subject or his/her legal guardian or caregiver.

  (4) Willingness and ability to cooperate with all programs of this study.

Exclusion Criteria:

- (1) Severe hepatic or renal insufficiency; (2) Targeted therapy before radiotherapy or PET/CT scan. (3)Renal function: serum creatinine less than or equal to the upper limit of the normal range;Liver function: bilirubin, AST(SGOT)/ALT(SGPT) less than or equal to the upper limit of the normal range.

(4) History of serious surgery in the last month. (5) Those who have participated in other clinical trials during the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess the sensitivity and specificity of using [18F]F-H3RESCA-3A12 and [68Ga]Ga-NOTA-3A12 for the diagnosis of metastatic gastric and pancreatic cancer | 90mins from time of injection
  In this study, we will first investigate the safety and feasibility of [18F]F-H3RESCA-3A12 and [68Ga]Ga-NOTA-3A12 in metastatic gastric and pancreatic cancers. The secondary goal of the clinical trial is to preliminary assess the sensitivity and specificity of using [18F]F-H3RESCA-3A12 or [68Ga]Ga-NOTA-3A12 PET/CT imaging for the diagnosis of metastatic gastric or pancreatic cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- PET Center, Huashan Hospital, Fudan University, Shanghai, China